CLINICAL TRIAL: NCT05250154
Title: Rheumatic Heart Disease Research and Screening in Nepal: A Feasibility Study
Status: Active, not recruiting | Type: Observational
Sponsor: University of Washington (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH); Fogarty International Center of the National Institute of Health (NIH)
Responsible Party: Principal Investigator, Nona Sotoodehnia, Associate Professor, School of Medicine, University of Washington
Other Study IDs: STUDY00005371; R34HL143279 (NIH); R21TW011108 (NIH)
Record Dates: First submitted 2021-10-18; First posted 2022-02-22 (Actual); Last update posted 2023-06-05 (Actual); Status verified 2023-06

CONDITIONS: Rheumatic Heart Disease
MeSH Terms: conditions — Rheumatic Heart Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Rheumatic Heart Disease (RHD) remains a significant public health problem in lower and middle-income countries, accounting for over 300,000 deaths world-wide. RHD is a sequela of Acute Rheumatic Fever (ARF) caused by Group A Streptococcus (GAS). Benzathine Penicillin Prophylaxis (BPP), through tri-weekly intramuscular injection of benzathine penicillin G, remains the mainstay of intervention to delay and prevent the sequelae among ARF and RHD patients by preventing repeat GAS infections. Two major obstacles exist to the optimal utilization of this effort. First, despite proven benefits, BPP adherence remains low. Unfortunately, there is very little knowledge on the factors associated with BPP adherence. Even in countries like Nepal, which has a nation-wide free BPP program serving about 6000 patients, there is absence of a robust system to prospectively track and study these patients. Second, largely because RHD is initially asymptomatic, only a fraction of those who would benefit are enrolled in BPP programs. There is a dearth of information and evidence on potentially high-yield approaches like the screening of first-degree relatives (FDRs) of RHD patients to identify asymptomatic, early-stage RHD patients who may benefit from BPP. The investigators will combine the resources and expertise at the University of Washington with those from existing partners at two leading Nepali hospitals (Manmohan Cardiothoracic Vascular and Transplant Center and Dhulikhel Hospital) to first create an easy to use, scalable, comprehensive electronic RHD registry and enroll BPP patients from these sites. In Aim 1, the investigators will examine whether patient socio-demographic, clinical, and health services-related characteristics are associated with BPP adherence. Investigators will use the BPP registry to collect important covariate information and adherence outcomes to address this aim. In Aim 2, investigators will determine the feasibility of screening FDRs of known RHD patients. Investigators will invite FDRs of known RHD patients (enrolled in the BPP registry) for echocardiographic screening for RHD. Investigators will assess the prevalence of RHD in these FDRs. This proposal harnesses one of the largest RHD patient pools in the world for establishing a robust RHD-related quality improvement and research platform that serves as a solid foundation for conducting larger epidemiologic, interventional, and implementation studies on RHD risk, prevention, and treatment.

ELIGIBILITY:
Inclusion Criteria:

* RHD patients

Exclusion Criteria:

-

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Registry of RHD patients
Sampling Method: Non-Probability Sample
Enrollment: 2438 (Actual)
Dates: Start 2018-08-27 (Actual); Primary Completion 2040-05-01 (Estimated); Study Completion 2040-05-01 (Estimated)

PRIMARY OUTCOMES:
Progression of rheumatic heart disease valve measured using standard imaging protocols | 20 years
  We will use standard imaging protocols to evaluate mitral, aortic, and tricuspid valves, which will allow analysis according to the World Heart Federation criteria for echocardiographic diagnosis of RHD among adults
Adherence to BPP measured using proportion of days covered. | 20 years
  The BPP clinic staff will enter information on injection every three weeks and will make a note of any clinical events during the preceding 3 weeks as reported by the patients. We will prospectively follow for one year all patients recruited in the first six weeks. At one year, we will assess the adherence to BPP. We will measure adherence using the proportion of days covered (PDC). PDC, a commonly used pharmacy quality measure for oral medications, has been adapted for injectable BPG in prior reports.

CONTACTS AND LOCATIONS:
Overall Officials: Nona Sotoodehnia, MD, MPH, Principal Investigator — University of Washington
Locations (1):
- Dhulikhel Hospital, Dhulikhel, Kavre, Nepal